CLINICAL TRIAL: NCT00656227
Title: A Double Blind, Placebo Controlled Randomised Trial to Investigate the Scar Improvement Efficacy of a Single Intradermal Application of RN1001 (Avotermin) in Subjects Undergoing Excision of Benign Head and Neck Naevi.
Brief Title: A Trial to Investigate Scar Improvement Efficacy of RN1001 (Avotermin) After Head and Neck Naevi Excision
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renovo (Industry)
Responsible Party: Dr Jim Bush, Renovo Clinical Trials Unit
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: RN1001-319-1008
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Nevus; Cicatrix
MeSH Terms: conditions — Nevus; Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Avotermin — Comparison of different dose levels (20ng, 50ng, 100ng or 200ng/100 ul) versus placebo

SUMMARY:
This trial will investigate whether four doses of RN1001 (20ng, 50ng, 100ng and 200ng) are efficacious in preventing or reducing the resultant scar, as compared to placebo, when applied intradermally to wound margins following excision of benign naevi situated on the head and neck.

DETAILED DESCRIPTION:
Male and female subjects (aged between 18-85 years) with one or more benign head & neck naevi will be invited to participate in the study.

Each patient will be randomised to a particular dose group, depending on the number of naevi suitable for excision. For example, patients with one excised naevi will receive either a dose of one of the concentrations of RN1001, or placebo. A patient with 2 excised naevi will receive an active dose, and placebo. Patients with 3 excised naevi will receive 2 active doses, plus placebo, and patient with four excised naevi will receive 3 active doses plus placebo.

Naevi will be excised using punch biopsy, and then closed with standard sutures. Following wound closure, the study drug (active RN1001 or placebo) will be administered via intradermal injection at a rate of 100ul per linear cm of wound margin.

Digital and film photography will be taken pre-dose and post dose (Day 0, day 14, day 28, Month 2, 3, 6 & 12, and thereafter at M24, M36, M48 & M60). Additionally, scar assessments (completed by Investigator, Research Nurse & Medical photographer) will be completed at follow up visits from Day 20 onwards. Silicone moulds of the scars will be taken at M6, M12 and then annually to M60.

Patients will be requested to complete a questionnaire to rate their scar expectations/assessment on a total of 5 occasions (screening, Day 0, Month 3, Month 6 & Month 12)

ELIGIBILITY:
Inclusion Criteria:

* Weight between 50 and 150kg and a body mass index within the permitted range for their height, using Quetelet's index-weight (kg)/height² (m). The permitted index is between 15-55.
* Subjects with one or more benign head and neck naevi which when measured are at least 3cm apart.
* Subjects who are aged 18-85 years.

Exclusion Criteria:

* Subjects who on examination have a naevus or naevi, which appear clinically suspicious of malignancy and therefore require specialist referral and treatment.
* Subjects who on direct questioning and physical examination have a history or evidence of hypertrophic or keloid scarring or tattoo(s) or previous scar(s) in the area to be excised.
* Subjects with a personal history of a bleeding disorder.
* Subjects with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of acute wounds or involves the areas to be examined in this trial.
* Subjects with any clinically significant medical condition that would impair wound healing including renal, hepatic, haematological, neurological or immune disease.
* Subjects with a history of clinically significant drug hypersensitivity to lignocaine or allergy to surgical dressings to be used in this trial.
* Subjects with any clinically significant abnormality following review of pre trial laboratory data and physical examination.
* Subjects who are taking, or have taken, any investigational drugs within the last 30 days, long term oral, topical or inhaled corticosteroid therapy and anti coagulant or anti platelet medication.
* Certain drugs are not excluded in this trial. These include OTC analgesics including paracetamol and codeine, vitamin and mineral supplements and OTC cold remedies containing paracetamol as the active ingredient.
* Subjects who are pregnant or who become pregnant up to and including Day 0. Subjects must use suitable forms of contraception during at least the first two months of the trial.
* Subjects who have previously had a positive result to the test for HIV antibodies, or who admit to belonging to a high-risk group.
* In the opinion of the Investigator, a subject who is not likely to complete the trial for whatever reason.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2004-04; Primary Completion 2007-07 (Actual); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Month 12 VAs - difference between active and placebo | 12 month

SECONDARY OUTCOMES:
VAS from the independent external panel | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MB ChB, Principal Investigator — Renovo Clinical Trials Unit
Locations (1):
- Renovo Clinical Trials Unit, Manchester, United Kingdom